CLINICAL TRIAL: NCT04314882
Title: The Danish National Survey of Diet and Physical Activity 2021-2024
Acronym: DANSDA
Status: Completed | Type: Observational
Sponsor: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Sisse Fagt, senior advisor, Technical University of Denmark
Other Study IDs: H-19033428
Record Dates: First submitted 2020-02-27; First posted 2020-03-19 (Actual); Last update posted 2025-05-02 (Actual); Status verified 2023-07

CONDITIONS: Diet Habit; Nutritional and Metabolic Disease; Lifestyle
Keywords: Diet; Nutrition; Physical activity; Lifestyle; Metabolic syndrome; Anthropometrics; Blood pressure; Pedometer-determined steps; BMI; Waist circumference; Metabolic health biomarkers
MeSH Terms: conditions — Feeding Behavior; Metabolic Diseases; Motor Activity; Metabolic Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Blood samples (whole blood, serum, plasma)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Danish National Survey of Diet and Physical Activity (DANSDA) 2021-23 is a nationally representative, cross-sectional survey of dietary and physical activity habits of 4-80 year-old Danes, and is carried out at the National Food Institute, Technical University of Denmark (DTU Food). DANSDA provides high quality, nationally representative data on diet, physical activity, smoking, alcohol and weight status in Denmark.

DETAILED DESCRIPTION:
The principal objective of DANSDA is to monitor dietary intake and physical activity in a representative sample of the Danish population aged 4-80 years, and provide data for surveillance of the food and nutrient intake and physical activity of the general population.

The survey is a nationally representative cross-sectional survey, which includes face-to-face interviews, anthropometric measurements, blood pressure measurement, blood sampling, 7-day web-based food diaries, and pedometer-determined physical activity which is recorded in 7-day web-based step diaries. In the interview socio-demographic details as well as lifestyle and health attitudes are recorded. Web-based food and step diaries are collected in the entire survey population of 4000 individuals, blood pressure is measured in 15-80 year-olds, and biological samples (blood) are collected in a subpopulation of approximately 1000 individuals aged 40-70 years. Biomarker of metabolic health are measured in a blood sample drawn after an overnight fast. The blood-based biomarkers (cholesterol, triglycerides, glucose), anthropometric data and blood pressure measurements are used to assess the prevalence of the metabolic syndrome (WHO definition) in 40-70 year-old Danes. Surplus blood samples are stored in a biobank for 30 years.

The data from the survey provide the evidence base to support work by the authorities to facilitate the adoption of healthier eating and physical activity behavior and reduce lifestyle-related diseases. Another objective is to provide detailed data on food consumption at the individual level, which enables food chemical exposure assessment and forms an essential part of food safety risk assessment. Furthermore, the data will be used to assess the environmental impact of the diet.

ELIGIBILITY:
Inclusion Criteria:

* Danish Citizen
* 4-80 years old
* Sufficient Danish language proficiency

Exclusion Criteria:

* Care home resident

Ages: 4 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The survey population consists of a nationally representative sample of 4-80-year-old Danes, randomly drawn from the Danish Civil Registration system.
Sampling Method: Probability Sample
Enrollment: 4224 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Dietary intake | Baseline
  Dietary intake is assessed by a 7-day web-based food diary.

SECONDARY OUTCOMES:
Physical activity | Baseline
  Physical activity is assessed by pedometer recordings over 7 days, measured as daily steps
Intakes of rare food products | Baseline
  Supplementary food frequency questionnaire (FFQ) focusing on foods consumed occasionally
Blood pressure | Baseline
  Average of three blood pressure measurements (systolic and diastolic blood pressure) using a validated blood pressure monitor, measured in mmHg. Measured among 15-80-year-olds.
Waist circumference | Baseline
  Waist circumference, measured in cm
Body mass index | Baseline
  Weight and height will be combined to report BMI in kg/m^2
Fasting glucose | Baseline
  Fasting glucose concentration in plasma, measured in mmol/l among 40-70-year-olds
Triglyceride | Baseline
  Plasma triglyceride concentration, measured in mmol/l among 40-70-year-olds
HDL cholesterol | Baseline
  Plasma HDL concentration, measured in mmol/l among 40-70-year-olds
Total cholesterol | Baseline
  Plasma total cholesterol concentration, measured in mmol/l among 40-70-year-olds
Metabolic syndrome score | Baseline
  Waist circumference, blood pressure, HDL cholesterol, triglycerides and fasting glucose will be combined to report metabolic syndrome score among 40-70-year-olds.
Socio-demographic background information through personal interview | Baseline
  Personal interview about socio-demographic background, lifestyle and health attitudes

CONTACTS AND LOCATIONS:
Overall Officials: Sisse Fagt, Principal Investigator — Technical University of Denmark
Locations (1):
- Technical University of Denmark, Copenhagen, Kgs Lyngby, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Survey home page — http://www.dansda.food.dtu.dk/